CLINICAL TRIAL: NCT06785662
Title: The Efficacy of Budesonide Nasal Irrigation in Allergic Rhinitis Patients: A Randomized, Controlled Trial.
Brief Title: Budesonide Irrigation in Allergic Rhinitis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Navarat Kasemsuk, Dr., Siriraj Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Si044/2022
Record Dates: First submitted 2025-01-13; First posted 2025-01-21 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: Allergic Rhinitis
Keywords: intranasal corticosteroid; budesonide nasal irrigation; Budesonide nasal spray; Allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Intervention Model Description: This trial will be reported according to CONSORT 2010 statement for randomized controlled trials. The enrolled participants were assigned a study code that was enclosed in a sealed envelope, prepared by personnel not involved in the research, and then randomly allocated into one of two groups using a computer-generated random permuted blocks design. The outcomes assessors were blinded to the randomization.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- The budesonide nasal irrigation group (Experimental): The participant in this group used a solution containing 1 milligram of budesonide mixed with 240 milliliters of normal saline in a squeeze bottle (Cleanoze®) for nasal irrigation. The procedure will be performed once daily while leaning slightly forward over a sink.
  Interventions: Drug: The budesonide nasal irrigation
- The budesonide nasal spray group (Active Comparator): The participant in this group used a nasal spray containing 64 micrograms of budesonide per spray, with two sprays per nostril administered twice daily (morning and evening).
  Interventions: Drug: The budesonide nasal spray

INTERVENTIONS:
Drug: The budesonide nasal irrigation — The participant in this group used a solution containing 1 milligram of budesonide mixed with 240 milliliters of normal saline in a squeeze bottle (Cleanoze®) for nasal irrigation. The procedure will be performed once daily while leaning slightly forward over a sink.
  Arms: The budesonide nasal irrigation group
Drug: The budesonide nasal spray — The participants in this group used a nasal spray containing 64 micrograms of budesonide per spray, with two sprays per nostril administered twice daily (morning and evening).
  Arms: The budesonide nasal spray group

SUMMARY:
Topical nasal steroids are significant therapeutic options for allergic rhinitis (AR). The distribution of intranasal steroid spray (INS) administration is less than that of irrigation. However, the available data on steroid nasal irrigation is limited. This article aims to evaluate the efficacy and adverse effects (AEs) of steroid irrigation in AR patients.

DETAILED DESCRIPTION:
Allergic rhinitis is a prevalent health problem found in Thai population, with various treatment approaches available, such as avoiding triggering allergens, using pharmacological treatments, receiving allergy immunotherapy, and going on a surgery.[1] Nowadays, the use of topical medications, particularly steroids, plays a crucial role in treating nasal and sinus conditions due to their anti-inflammatory properties. Normally, steroids can be administered through diverse methods including nasal sprays, drops, and irrigation. The general guidelines for treating allergic rhinitis or chronic sinusitis typically emphasized the use of topical nasal steroids, particularly in spray form.[2, 3] Other forms of drug administration are generally considered alternative options. However, studies have shown that the distribution of medication via nasal spray is inferior to that of other delivery methods, including nasal irrigation. Most of the medication is concentrated in the anterior portion of the nasal cavity, particularly the nasal vestibule, with limited distribution to the inferior turbinate, superior turbinate, sphenoethmoidal recess, and superior olfactory cleft, compared to nasal irrigation. Therefore, the administration of topical steroids by nasal irrigation may serve as an alternative topical steroid delivery method.[4] Previous studies have mentioned the use of steroid nasal irrigation, primarily in patients with post-endoscopic sinus surgery for chronic sinusitis.[5-17] Additionally, there have been studies addressing its application in conditions such as allergic fungal rhinitis, acute sinusitis in children, and post-operative patients following septoplasty.[18, 19] The use of steroid nasal irrigation for treating allergic rhinitis has been scarcely discussed, and there is limited data available. One study investigated the use of budesonide nasal irrigation compared to normal saline nasal irrigation in patients with allergic rhinitis. The results showed that the Sinonasal Outcome Test-22 (SNOT-22) score and Visual Analog Scale (VAS) scores in the budesonide nasal irrigation group were significantly superior than those in the saline irrigation group.[20] However, there have been no studies conducted on patients with allergic rhinitis where nasal spray treatment was insufficient to control the symptoms of nasal inflammation. Additionally, no comparative studies between different drug administration techniques have been carried out.

This study aims to evaluate the efficacy of budesonide nasal irrigation in patients with allergic rhinitis, where the use of nasal steroid spray alone was insufficient to control nasal inflammation and required dosage adjustment. We hypothesized that administering steroids via nasal irrigation would improve drug distribution, leading to better outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18-60 years diagnosed with perennial allergic rhinitis based on ARIA guidelines, who have previously consistently used intranasal corticosteroids for at least 2 weeks with inadequate control of nasal inflammation defined by a VAS score of ≥5 out of 10 and requiring dosage adjustment. Noted that proper technique should have been confirmed through retrospective questioning.

Exclusion Criteria:

* Those with a history of sinus surgery, nasal or sinus tumors (including polyps), significant deviated nasal septum causing symptoms, oral corticosteroid uses for any indication, immunodeficiency, pregnancy, breastfeeding, or suspected fungal sinusitis indicated by ischemic nasal tissue, fungal masses, bone erosion, or calcifications on imaging were excluded. Participants would be withdrawn if severe complications arise from the use of topical budesonide.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-02-12 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Total Nasal Symptom Score (TNSS) | Follow-up visits were scheduled at 2 and 4 weeks after starting treatment.
  Full Name: Total Nasal Symptom Score Scale Range: 0 to 12 Scoring Interpretation: Higher scores indicate a worse outcome
  Each symptom is rated by the participant on a scale (0 to 3), based on severity:
  0: No symptoms
  1. Mild symptoms (present but not bothersome)
  2. Moderate symptoms (noticeable and somewhat bothersome)
  3. Severe symptoms (very bothersome and interfering with daily activities)

SECONDARY OUTCOMES:
Postnasal Drip Symptom Score (PND) | Follow-up visits were scheduled at 2 and 4 weeks after starting treatment.
  Postnasal Drip Symptom Score (PND) determines the severity of post nasal drip sensation
  Full Name: Postnasal Drip Symptom Score Scale Range: 0 to 3 Scoring Interpretation: Higher scores indicate a worse outcome. The PND focuses specifically on the severity of postnasal drip symptoms, with scores representing none (0), mild (1), moderate (2), or severe (3) symptoms.
Rhinoconjunctivitis Quality of Life Questionnaire (RCQ-36) | Follow-up visits were scheduled at 2 and 4 weeks after starting treatment.
  Rhinoconjunctivitis Quality of Life Questionnaire (RCQ-36) determine disease-specific quality of life
  Full Name: Rhinoconjunctivitis Quality of Life Questionnaire - 36 Items Scale Range: 0 to 6 for each item, summing up to a total score. Scoring Interpretation: Higher scores indicate a worse outcome. This questionnaire assesses the impact of rhinoconjunctivitis symptoms on quality of life, covering domains such as sleep, activities, emotional well-being, and social functioning.
Peak Nasal Inspiratory Flow (PNIF) | Follow-up visits were scheduled at 2 and 4 weeks after starting treatment.
  Peak Nasal Inspiratory Flow (PNIF) is an objective measurement to determine nasal patency
  Full Name: Peak Nasal Inspiratory Flow Scale Range: Measured in liters per minute (L/min); there is no fixed maximum value, as it depends on individual physiology.
  Scoring Interpretation: Higher values indicate a better outcome. PNIF measures the maximum airflow through the nasal passages during inspiration and is used as an objective measure of nasal patency (openness).
Adverse events | Follow-up visits were scheduled at 2 and 4 weeks after starting treatment.
  All adverse events occurred during the usage of budesonide nasal irrigation were reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Siriraj Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No